CLINICAL TRIAL: NCT05042349
Title: Pregnant Elite Athletes and Pregnant Women Exercising With Moderate Intensity
Status: Withdrawn | Type: Observational
Why Stopped: no funding
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: 125635
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Body Image; Physical Activity; Exercise; Energy Intake; Nutritional Status; Pregnancy Related; Fetus Risk; Blood Flow; Body Temperature
Keywords: Pregnancy; Elite athlete; Fetus; Physical health; Mental health
MeSH Terms: conditions — Motor Activity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Elite athletes: Pregnant female elite athletes
- Controls: Moderately physical active pregnant females
- Sponsors: Sponsors of the athletes
- Coaches/tema leaders: Coaches or team leaders of the atheltes

SUMMARY:
The aim of this study is to 1. register possible changes to uteroplacental circulation in relation to physical tests, 2. to register energy and nutritional intake, relationship towards the body during pregnancy and during the early period after giving birth, 3. register the experience of guidance given related to exercise, nutrition, and recovery, 4. register elite athletes' experience of combining the role of being a mom and an elite athlete, and 5. register attitudes and reactions from the support system when it comes to being an elite athlete and being pregnant. Material and method: 30 pregnant female elite athletes and 30 moderately physically active pregnant women will be recruited for the completion of physical testing and questionnaires and questionnaires only, respectively. 20 national team leaders/coaches and 10 sponsors will be recruited for a semi-structured interview about attitudes, reactions and guidance towards athletes who become pregnant and still wish to continue their career as an athlete after pregnancy.

DETAILED DESCRIPTION:
The aim of this study is to 1. register possible changes to uteroplacental circulation in relation to physical tests, 2. to register energy and nutritional intake, relationship towards the body during pregnancy and during the early period after giving birth, 3. register the experience of guidance given related to exercise, nutrition, and recovery, 4. register elite athletes' experience of combining the role of being a mom and an elite athlete, and 5. register attitudes and reactions from the support system when it comes to being an elite athlete and being pregnant. Material and method: It is expected that we can include 30 pregnant female elite athletes for the physiological testing who also will complete the questionnaires included in the study. In addition, 30 moderately physically active pregnant women will be recruited for the completion of the questionnaires only. Both groups answer questions related to exercise, pregnancy related issues, nutrition and their relationship towards their body. To obtain enough participants, data collection will continue for five years. During the same period, 20 national team leaders/coaches and 10 sponsors will be recruited for a semi-structured interview. The physiological testing will be conducted during the 23-29th week of pregnancy. The athletes will conduct a running test and resistance tests in the lab. The following measures will be registered: pulsatility index (PI) and volume blood flow in both uterine arteries, 2. the fetus' pulsatility index (PI) in the umbilical cord artery and heart rate frequency, 3. body temperature, heart rate, blood pressure and saturation in the mother during rest and during physical exertion. Data on gestational development and birth will be collected based on information given by the participant herself and by birth records and health records. Coaches/leaders and sponsors will in their interview, answer to questions related to attitudes, reactions and guidance of athletes who become pregnant and still wish to continue their career as an athlete after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Athletes: pregnant female pregnant elite athletes at a recruiting team, junior or senior, who represent athletes within endurance, weight sensitive, ball sports, and technical sports.
* Controls/reference group: pregnant females who are moderately physically active.
* For both groups: age 18-40 år.

Exclusion Criteria:

* Known illness or disease, which defines their pregnancy as a high-risk pregnancy
* Age >40 years old.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants need to be female only for the athletes and the control/reference group. For the sponsors, coaches and team leaders, there are no gender specifications or inclusion criteria.
Study Population: The sample represents 1. pregnant female elite athletes, 2. pregnant females who are only moderately physically active, 3. the athletes sponsors, 4. the athletes coach/team leader.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Exercise | 5 minutes
  Self-developed questions about exercise volume before, during, and after pregnancy. Participants respond to open ended questions and questions with yes/no and multiple response options.
Fertility and pregnancy related issues | 5 minutes
  Participants respond to open ended questions and questions with yes/no and multiple response options.
Nutrition | 5 minutes
  Questionnaire. Four days of dietary registration during, where participants respond both to questions with Likert scales, YES/NO, and multiple response options, 1st, 2nd, 3rd trimester, and 3 months after delivery.

SECONDARY OUTCOMES:
Pulsatility index | 15 minutes
  Ultrasound
Volume blood flow | 5 minutes
  Ultrasound
Heart rate frequency | 5 minutes
  Heart rate monitor
Body temperature | 5 minutes
  Thermometer
Blood pressure | 10 minutes
  Sphygmomanometer
Attitudes, reactions and guidance of athletes who become pregnant and still wish to continue their career as an athlete after pregnancy | 5 minutes
  Participants respond to open ended questions and questions with yes/no and multiple response options.
Satisfaction with life | 1 minute
  Satisfaction with life scale. 5 items answered on a 7-point Likert scale, where higher sum score indicates higher satisfaction with life
Beck's Depression Inventory (BDI-IA) | 1 minute
  Questionnaire where five questions are answered to on a 6-point Likert scale, with higher score indocates higher level of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, PhD, Principal Investigator — The Norwegian School of Sport Sciences
Locations (1):
- The Norwegian school of sport sciences, Oslo, Norway